CLINICAL TRIAL: NCT04971525
Title: An Observational European Multi-database Linkage Study to Quantify Malignancy Rates in Crohn's Disease Patients With Complex Perianal Fistula Treated With Darvadstrocel
Brief Title: A Study to Check How Often People Treated With Darvadstrocel for Crohn's Disease Are Diagnosed With Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Sponsors decision
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alofisel-5005
Record Dates: First submitted 2021-07-19; First posted 2021-07-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease; Complex Perianal Fistula
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Darvadstrocel Cohort: Participants diagnosed with CPF-CD, who administered at least one dose of darvadstrocel in fistula tract tissue under surgical environment will be observed.
- Matched Control Cohort: Standard of Care (SoC): Participants diagnosed with CPF-CD with no history of administration of darvadstrocel, matched age at index date (within 3 years), sex and if feasible, complex perianal fistula (CPF) diagnosis (within 1 year) to individuals in the darvadstrocel cohort who received the alternative Standard of Care (SoC), which varies from country to country and according to local centre expertise will be observed.

SUMMARY:
The main aim is to learn about the risk of cancer after treatment with darvadstrocel compared to other standards of care in people with Crohn's Disease (CD).

In this study, the study doctors will review each participant's past medical records. This study is about collecting existing information only; participants will not receive treatment or need to visit a study doctor during this study.

DETAILED DESCRIPTION:
This is a retrospective, non-interventional study of participants with complex perianal fistula in Crohn's disease (CPF-CD). This study will assess tumorigenicity risk and all-cause and cancer-specific mortality in participants with darvadstrocel.

The study will enroll approximately 5850 participants. Data will be collected retrospectively from European secondary data sources. Participants will be assigned to two cohorts:

* Darvadstrocel cohort
* Matched control cohort: Alternate SoC.

This multi-center trial will be conducted in France, Germany, Netherlands, and Spain. The overall duration of the study will be approximately 96 months, including index period (the time in which eligible participants are included in the study) and 12 months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Darvadstrocel cohort 1. Participants will be included in the darvadstrocel cohort if they have at least one record of prescription/dispensation/administration of darvadstrocel at some point during the study period.

Comparator cohort

1. A comparator cohort of controls (matched control cohort) will be composed of participants with CD and PF randomly selected from a pool of eligible participants with no history of administration of darvadstrocel.

Exclusion Criteria:

1. Has less than 12 months of uninterrupted data within country-specific data source prior to index date.
2. Has not meet quality indicators for country-specific data source (if applicable).
3. Has diagnosis of cancer prior different from non-melanoma skin cancer to index date. This will minimise the misclassification of prevalent or metastatic cancer as incident cases for the analysis of the study objectives.
4. Has diagnosis of ulcerative colitis at any point during the study period and medical history period. This will avoid potential ascertainment bias as there is currently no gold standard for differential diagnosis in IBD. Approximately 5 percent (%) to 15% of cases do not meet strict criteria for either ulcerative colitis (UC) or CD and in up to 14% of participants classified as UC and CD, the diagnosis changes over time.
5. Has record of proctectomy or colectomy prior to index date. Proctectomy and colectomy are considered "last chance" surgery options for anal fistulas or other complications of CD. These participants are not the target population for darvadstrocel. They would not be eligible for darvadstrocel administration and loss of their gastrointestinal tract would affect the risk of colorectal cancer; the most common cancer associated with CD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with CPF-CD who have been administered at least one dose of darvadstrocel and participants with CD and perianal fistula (PF) and no history of administration of darvadstrocel.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Malignancies Among Participants With CPF-CD | Up to Month 96
  Incidence rate of malignancies will be calculated as the number of newly observed cases divided by the person-years of follow-up during that period.
Cumulative Incidence of Malignancies Among Participants With CPF-CD | Up to Month 96
  Cumulative incidence rate within a period will be calculated as the ratio of newly observed cases divided by the population at risk during that period.

SECONDARY OUTCOMES:
All-cause Mortality Rate Among Participants With CPF-CD | Up to Month 96
Cancer-specific Mortality Rate Among Participants With CPF-CD | Up to Month 96
Number of Participants With Anal Fistula Surgery | Up to Month 96
Number of Participants With Colorectal Surgery | Up to Month 96
  Colorectal surgery such as colectomy and proctectomy modify colorectal cancer risk. Colorectal surgery will be identified using procedure codes specific to each country-specific data source.
Number of Participants With CPF-CD Characterized by Pharmacological Therapies | Up to Month 96
  Thiopurines and methotrexate have been found to increase the risk of lymphoma and skin cancer. These drugs will be identified in outpatient prescription data using Anatomical Therapeutic Chemical (ATC) codes. In the case of in-hospital administered drugs, such as anti-tumour necrosis factor's (anti-TNF) and biologics, drugs will be defined using relevant ATC codes and/or procedure codes available in the hospital records.
Number of Participants With Comorbidities | Up to Month 96
  Comorbidities will be identified using International Classification of Diseases 10th revision (ICD-10 codes) (or country specific modifications) within hospital settings in each country-specific data source.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- 1. Système National des Données de Santé (SNDS), Charenton-le-Pont, France
- Institut für angewandte Gesundheitsforschung Berlin (InGef), Berlin, Germany
- PHARMO, Utrecht, Netherlands
- Estudio Nacional en Enfermedad Inflamatoria intestinal sobre Determinantes genéticos y Ambientales (ENEIDA), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/60f88e78f883ca001e82d35e